CLINICAL TRIAL: NCT06472271
Title: Colistin in Neonatal ICU Patients With Gram Negative Resistant Infection: Dosage Personalization Approach
Brief Title: Colistin Dosage Prsonalization Approach
Status: Recruiting | Type: Observational
Sponsor: Mahmoud I Mostafa (Other)
Responsible Party: Sponsor-Investigator, Mahmoud I Mostafa, Lecturer at pharmacy practice department, Helwan University
Organization: Helwan University (Other)
Other Study IDs: colistin in neonates
Record Dates: First submitted 2024-06-18; First posted 2024-06-25 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Colistin Adverse Reaction
MeSH Terms: interventions — Colistin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 21 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Conventional initial dose: Colistin 5mg/kg/day
  Interventions: Drug: Polymyxin e
- High initial dose: Colistin 7.5mg/kg/day
  Interventions: Drug: Polymyxin e

INTERVENTIONS:
Drug: Polymyxin e — Increased starting colistin dose
  Other Names: Colistin

SUMMARY:
A few studies have evaluated higher doses or the administration or a loading dose, which is routine in adults, in pediatric patients, and reported improved colistin exposure without an increased risk of nephrotoxicity The main questions it aims to answer are What is the optimal dosing strategies of intravenous colistin for the treatment of multidrug-resistant gram-negative bacterial infections in preterm neonates? What is the incidence of AKI? What is the factors increasing AKI incidence? A single center retrospective and comparative study, cohort study compare low dose 5 mg/kg/day versus 7.5mg/kg/day

DETAILED DESCRIPTION:
Retrospective study to measure safety and efficacy of colistin conventional dose versus high dose then prospective design to measure pharmacokinetics parameter of both doses to design optimal dose

ELIGIBILITY:
Inclusion Criteria:

* Neonates aged between (0-30 days) born before 37 weeks
* Critically ill patients with nosocomial infection with proven culture-resistant gram-negative bacteria.
* Neonates who are indicated for colistin and started colistin therapy for at least 48 hr.

Exclusion Criteria:

* Serum creatinine ≥1.5 baseline before colistin
* Received colistin before NICU stay
* Administration of concurrent nephrotoxic drugs including amphotericin, gentamicin, or amikacin.
* Major congenital anomalies or with previous renal impairment.

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm, critically-ill, neonates diagnosed with resistant gram-negative infections
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Clinical response | 21 days
  Resolving signs and symptoms with normalized acute phase reactants in clinical septic patients

SECONDARY OUTCOMES:
Microbiological clearance | 21 days
  Negative culture results following Colistin therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo univrsity Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided